CLINICAL TRIAL: NCT06318988
Title: An Observational, Prospective Study to Assess the Outcomes of Different Treatment Options in Patients With Chronic Venous Disease in Belgium
Brief Title: Outcomes of Different Treatment Options in Chronic Venous Disease
Acronym: VOS
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S67030
Record Dates: First submitted 2024-02-29; First posted 2024-03-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Chronic Venous Disease
MeSH Terms: interventions — Polidocanol; Diosmin; troxerutin; Antistax; Stockings, Compression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conservative: compression therapy, and oral or topical venoactive drugs
  Interventions: Drug: Daflon; Device: Compression stocking
- invasive: sclerotherapy, foamsclerotherapy, open surgery, endovenous thermal ablation
  Interventions: Procedure: Radiofrequency ablation using Closure fast; Procedure: Aethoxysclerol

INTERVENTIONS:
Procedure: Radiofrequency ablation using Closure fast — Thermal ablation technique
  Other Names: Laserablation using laser fiber
  Groups: invasive
Procedure: Aethoxysclerol — sclero-or foamsclerose
  Other Names: polidocanol
  Groups: invasive
Drug: Daflon — Venoactive drugs
  Other Names: Venoruton; Antistax
  Groups: conservative
Device: Compression stocking — Compression
  Groups: conservative

SUMMARY:
This study aims to describe conservative and invasive treatments for patients with chronic venous disease (CVD) in Belgium, and their association with clinical and patient-reported outcomes during a follow-up of 24 months.

DETAILED DESCRIPTION:
This study is an observational, prospective, multicentre study to assess the effectiveness of conservative and invasive treatments in patients with CVD in Belgium. The inclusion period of the study will last 6 months. Patients will be followed until 2 years after inclusion into the study.

During the inclusion period, after confirmation of eligibility, patients with CVD diagnosed by the General Practitioner (GP) and requiring a treatment will be invited to participate in the study. About 140 GPs across Belgium will be included in the study. During the first visit, a treatment strategy will be proposed to the patient by the GP. The treatment can be conservative or invasive, depending on the severity of the disease. Patients awaiting invasive treatment may receive conservative treatment to alleviate symptoms. The choice of treatment modality is left to the discretion of the treating physician, in agreement with the patient and according to local policies. As this is an observational study, there will be no interference in the choice of treatment, and no restrictions will be imposed.

ELIGIBILITY:
Inclusion Criteria:

* Patient visiting a GP with complaints related to CVD,

* Patient receiving the diagnosis of CVD from the GP during the V0, according to international guidelines and made on a clinical basis,
* Patient requiring and agreeing to receive conservative or invasive treatment,
* French or Dutch speaking patient,
* Patient signed informed consent and agrees to take part in the study and follow-up.

Exclusion Criteria:

* Patient with coagulation disorders such as thrombophilia and/or taking anticoagulation drugs,
* Pregnant or breastfeeding patient,
* Patient with severe Peripheral Arterial Occlusive Disease (POAD), with Ankle Brachial Index (ABI) < 0.8,
* Patient with malignancy,
* Patient with neurological disorder or dementia,
* Patients taking regular treatment for CVD 3 months prior to inclusion (except painkillers or anti-inflammatory drugs if taken for reasons other than CVD),
* Patient in any other clinical study for any pharmaceutical product within 4 weeks preceding study inclusion,
* Patient with any comorbidity or situation preventing a follow-up of 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic venous disease who did not receive any dedicated treatment for CVD 3 months prior to inclusion
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Chronic Venous Insufficiency QOL questionnaire- 20 (CIVIQ-20) score | baseline to 12 weeks
  Chronic Venous Insufficiency QOL questionnaire-20 score, min 20 max 100, higher means worse outcome

SECONDARY OUTCOMES:
Intervention as secondary/add-on treatment | month 24
  Proportion of patients who received an intervention as secondary/add-on treatment to conservative treatment
The change in the Chronic Venous Insufficiency QOL questionnaire-20 score (CIVIQ-20) | through study completion, an average of 2 years
  The change in the CIVIQ-20 over time; min 20 max 100, higher means worse outcome
The change in the clinical part of the Clinical, Etiological, Anatomical and Pathophysiological classification (CEAP classification) | through study completion, an average of 2 years
  The change in the clinical part of the CEAP classification over time, min C0, max C6, higher means worse outcome
The change in the revised Venous Clinical Severity Score (rVCSS) | through study completion, an average of 2 years
  The change in the rVCSS over time; min 0 max 30, higher means worse outcome
The change in the symptoms, recorded with a questionnaire | through study completion, an average of 2 years
  The change in the symptomatology over time, recorded with a questionnaire
The change in satisfaction score | through study completion, an average of 2 years
  The change in satisfaction score over time, min 0, max 10; higher means better outcome
Adverse Events (AEs). | month 24
  Number and proportion of patients with Adverse Events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Thomis, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven